CLINICAL TRIAL: NCT02568072
Title: Increased Left Ventricular Trabeculation in Athletes - a Marker of Left Ventricular Non-compaction or a Physiological Epiphenomenon of Increased Cardiac Preload?
Brief Title: Training-induced Increased Left Ventricular Trabeculation
Acronym: MARATHON
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: St. Bartholomew's Hospital (Other); Cardiac Risk in the Young (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 15.0035; FS/15/27/31465 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2015-09-28; First posted 2015-10-05 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Athletes Heart; Left Ventricular Hypertrabeculation
Keywords: exercise; cardiac remodelling; left ventricular non-compaction cardiomyopathy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples. Urine samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will expand on research conducted by the investigators' group, where the investigators have demonstrated increased LV trabeculation, satisfying currently existing criteria for LV Non-Compaction Cardiomyopathy (LVNC), in groups exposed to high cardiac workloads. To the investigators' knowledge, this will be the first prospective study aiming to demonstrate a direct relationship between high levels of exercise and increased LV trabeculation. This study may add weight to the theory that this entity currently described as LVNC, is a morphological epiphenomenon common to many distinct myocardial remodeling processes associated with increased cardiac preload and afterload and may better define normal adaptive increases in LV trabeculation.

DETAILED DESCRIPTION:
Background of Left Ventricular Non-Compaction Cardiomyopathy Left Ventricular Non-Compaction Cardiomyopathy (LVNC) is a myocardial disorder defined by increased left ventricular (LV) trabeculation and intertrabecular recesses communicating with the LV cavity. The condition is associated with progressive heart failure, systemic thromboembolism and a predilection to fatal ventricular arrhythmia and sudden cardiac death. However, a large proportion of affected individuals may be asymptomatic. One cohort study demonstrated 28% of detected cases of LVNC were asymptomatic, with the majority being identified through family screening. It must be emphasized that currently there is no diagnostic tool, neither genetic nor imaging, that can categorically identify an individual as having LVNC or not. This lack of a 'gold standard' makes the description of increased left ventricular trabeculation difficult, creating a tendency to apply a diagnostic label of LVNC inappropriately.

Traditional thought has been that LVNC results from arrest of the normal trabecular regression and myocardial compaction that occurs during embryological development. However, this concept is challenged by reported cases of 'acquired' LVNC, where serial echocardiograms have demonstrated a transition from a normal endocardial appearance to a hypertrabeculated LVNC phenotype. Whether this is a delayed presentation of a genetically heterogeneous cardiomyopathy or a morphological epiphenomenon shared by many phenotypically distinct cardiomyopathies, remains unknown. This irresolution is exemplified by international discordance, with the American Heart Association classifying LVNC as a genetic cardiomyopathy and the European Society of Cardiology and World Health Organisation taking the view that LVNC remains an 'unclassified cardiomyopathy'.

In the absence of congenital heart disease, LVNC was thought to be an extremely rare condition with a prevalence between 0.05% and 0.24%. Technical advances in echocardiography, largely second harmonic imaging, have led to improvement in LV apex and lateral wall visualization, which has dramatically increased the frequency of detection in the last 20 years.

Limitations in current diagnostic criteria At present, various diagnostic criteria exist entirely based on morphological findings on echocardiography or magnetic resonance imaging (MRI). All of these criteria have limitations in that they are generated from small patient cohorts, have substantial inter-observer variability and poor correlation between them. This is perhaps not surprising as they all measure different parameters in different echo planes and during different phases of the cardiac cycle.

In a study by Kohli et al, 24% of heart failure patients had at least one of three diagnostic echocardiography criteria for LVNC (Chin 19%, Jenni 15%, Stollberger 13%), as well as 8% of healthy controls, most of whom were of black ethnicity. Only 7% fulfilled all three criteria, indicating the relatively poor concordance between these criteria. These studies highlight the concern that echocardiographic criteria are too sensitive and lack specificity, particularly in black individuals, resulting in over-diagnosis of LVNC.

Whilst MRI has advantages over echocardiography in tissue characterisation, superior contrast-to-noise and signal-to-noise ratio and greater ability to visualize the cardiac apex, CMR criteria for the identification of LVNC suffer the same limitations as for echocardiography. When applying CMR criteria from Petersen et al, a recent population-based prospective multi-ethnic cohort study identified 25.7% of a low-risk 'healthy' population meeting criteria for LVNC.

Currently, application of imaging-based criteria for diagnosis to low risk populations creates a considerable burden of anxiety, potential loss of opportunity/earnings, unnecessary investigations and clinical follow-up, with their associated costs to the National Health Service. There is a considerable need in this area to evaluate what cardiac imaging criteria contribute to the diagnosis of LVNC. Indeed, some propose integration of clinical criteria including malignant arrhythmias, thromboembolic events, neuromuscular disorders and family history of LVNC into a diagnostic algorithm, though none currently exist.

Influence of ethnicity in cardiac remodeling and pilot data Racial differences in cardiac remodeling have previously been described with respect to cardiac hypertrophy. Athletes develop physiological increases in LV wall thickness and cavity size in an adaptive response to high cardiac preload and afterload. This response is exaggerated in black athletes. For the purposes of this study, black ethnicity will be defined as a person of African or African-Caribbean origin. In a study comparing highly trained male athletes, 18% of black athletes exhibited left ventricular hypertrophy (LVH), as defined as an LV wall thickness of >12mm, compared with only 4% of white athletes (p<0.001)13.

The investigators' group has shown that athletes also display a higher prevalence of increased LV trabeculation compared with controls (18.3% vs 7.0%; p < 0.0001) with 8.1% of athletes fulfilling conventional echocardiographic criteria for LVNC. As with LVH, this difference in LV hypertrabeculation appears to be exaggerated in black athletes as compared to white athletes (28.8% vs 16.3%; p = 0.002).

The investigators' group has also investigated the presence of increased LV trabeculation in a population of sickle cell anaemia patients. Chronic anaemia of sickle cell disease is associated with an increased LV preload and high cardiac output. The investigators found increased LV trabeculation in 28% of sickle cell anaemia patients as compared with 12% of asymptomatic healthy black controls. 8% of sickle cell anaemia patients fulfilled both Chin and Jenni criteria for LVNC.

These studies have limitations in their cross-sectional design and therefore a relationship of temporal causality between increased cardiac preload and the development of increased LV trabeculations could not be established.

This led the investigators' group to conduct a longitudinal cohort study utilizing pregnancy as a model of increasing cardiac preload and observing the effects on LV trabeculation. During pregnancy, at 28-36 weeks gestation, in increase in LV trabeculation was seen in 25.4%, having demonstrated normal myocardium at baseline. Moreover, 7.8% of women fulfilled Chin and Jenni criteria for LVNC. In addition, black women appeared to demonstrate a higher prevalence of increased LV trabeculation as compared with white women (46% vs. 13%; p = 0.0003).

With this proposed study the investigators aim to be the first to demonstrate that LV hypertrabeculation can be induced with athletic training in individuals with structurally normal hearts and that this will return to baseline after de-training. Although the population sampled will be a healthy cohort, the implications of the investigators' findings would resonate throughout the cardiac imaging community and fundamentally change perspective on the clinical detection of increased left ventricular trabeculation. The investigators aim to go further than before and compare echocardiographic and CMR measurements of left ventricular trabeculation and investigate whether a positive correlation exists between improvement in cardiopulmonary performance and extent of de novo LV hypertrabeculation. The project will also enable the assessment of the impact of gender on the development of LV trabeculation.

Should the investigators' hypothesis prove correct, this would potentially avoid inappropriate diagnostic labelling, unnecessary anxiety, investigations, treatment, follow up and family screening. This study may strongly emphasize the need for more robust diagnostic criteria for the diagnosis of LVNC.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic and normotensive sedentary individuals (≤2 hours/week of physical activity) aged 18-35 years

Exclusion Criteria:

1. Hypertension;
2. Previous cardiac history;
3. Symptoms suggestive of cardiac disease;
4. Use of anabolic steroids;
5. Use of performance enhancing drugs;
6. Abnormal ECG (As defined by the proposed refined ECG screening criteria for black and white athletes published by the Investigators' group)
7. Left ventricular hypertrophy >15 mm in males and >12 mm in females;
8. Significant valvular heart disease or intra-cardiac shunt on echocardiography
9. Individuals with contraindications to cardiac MRI scanning
10. Pregnant or breastfeeding women.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants running first marathon event in Virgin London Marathon 2016.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sharma, MD FRCP FESC, Principal Investigator — St George's, University of London
Locations (1):
- Barts Heart Centre, London, United Kingdom

REFERENCES:
- See also: Participant information website — https://sites.google.com/site/firsttimemarathonstudy/

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: 120 subjects recruited into study. 18-35 years old and had never run a marathon distance previously. Individuals were excluded if they had pre-existing cardiovascular disease during preliminary investigations or contraindication to cardiac magnetic resonance (CMR).
Period: Overall Study
Arm/Group | Study Group
Started | 120
Completed | 68
Not Completed | 52
Not completed — Unavailable for appointment | 23
Not completed — Unable to contact | 3
Not completed — Diagnosis of Long QT Syndrome | 1
Not completed — Withdrawal by Subject | 1
Not completed — Sustained injury, marathon not run | 24

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 36
Region of Enrollment [Number; unit: participants]
  United Kingdom | 68

OUTCOME MEASURES:

1. Primary Outcome: Thickness of Compacted Myocardial Tissue (cm)
Description: Measured on echocardiography and cardiac magnetic resonance:
  1. Echocardiographic measure of compacted myocardial tissue (systole) - Jenni Compacted layer measurement (cm)
  2. Cardiac magnetic resonance measure of compacted myocardial tissue (diastole) - Petersen Compacted layer measurement (cm)
Time Frame: Baseline and 7 months
Population: One subject did not undergo cardiac magnetic resonance imaging post marathon due to first trimester pregnancy
  68 Participants underwent the "Jenni Compacted layer measurement (cm)" and 67 Participants underwent the "Petersen Compacted layer measurement (cm)"
Measure: Median (Inter-Quartile Range); unit: cm
Groups:
- Baseline: Study participants with places in the 2016 London Marathon assessed prior to training
- 7 Months: Study participants evaluated after completing the 2016 London Marathon
Arm/Group | Baseline | 7 Months
Number analyzed (Participants) | 68 | 67
cm
  Petersen Compacted layer measurement (cm) | 0.53 [0.45 to 0.63] | 0.56 [0.48 to 0.64]
  Jenni Compacted layer measurement (cm) | 0.8 [0.7 to 1.0] | 0.85 [0.7 to 1.0]
Statistical Analysis 1: Comparison: Baseline vs 7 Months; Test type: Superiority; p = 0.44, t-test, 2 sided

2. Primary Outcome: Thickness of Non-compacted Myocardial Tissue (cm)
Description: Measured on echocardiography and cardiac magnetic resonance:
  1. Echocardiographic measure of non-compacted myocardial tissue (systole) - Jenni Non-Compacted layer measurement (cm)
  2. Cardiac magnetic resonance measure of non-compacted myocardial tissue (diastole) - Petersen Non-Compacted layer measurement (cm)
Time Frame: Baseline and 7 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Baseline | 7 Months
Number analyzed (Participants) | 68 | 67
cm
  Petersen Non-Compacted layer measurement (cm) | 0.65 [0.44 to 0.84] | 0.58 [0.43 to 0.73]
  Jenni Non-Compacted layer measurement (cm) | 0.8 [0.5 to 1.0] | 0.8 [0.6 to 1.0]
Statistical Analysis 1: Comparison: Baseline vs 7 Months; Test type: Superiority; p = 0.71, t-test, 2 sided

3. Primary Outcome: Myocardial Fractal Dimension
Description: Measured on cardiac magnetic resonance, dimensionless unit and measure of endomyocardial boarder complexity. The higher the value the greater the endocardial boarder complexity and therefore the more trabeculation.
  Two measurements were made:
  1. Captur et al. Global mean left ventricular fractal dimension
  2. Captur et al. Maximum apical fractal dimension
  These values are between 1 and 2. Binarisation eliminates pixel detail originating from the blood pool. The edge image is covered by a series of grids. The minimum size is set to 2 pixels. The maximum size of the grid series is dictated by the dimensions of the bounding box, referring to the smallest rectangle that encloses the foreground pixels. Through the implementation of this 2D box-counting approach, a fractal output of between 1 and 2 is expected. The log-lot plot (e) produces a good fit using linear regression and yields a gradient equivalent to - FD (1.363).
Time Frame: Baseline and 7 months
Population: One subject did not undergo cardiac magnetic resonance imaging post marathon due to first trimester pregnancy
  67 Participants underwent the "Fractal Dimension analysis" with paired results at baseline and at 7 months.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Baseline | 7 Months
Number analyzed (Participants) | 68 | 67
unitless
  Captur et al. Global mean left ventricular fractal dimension | 1.20 (0.06) | 1.19 (0.05)
  Captur et al. Maximum apical fractal dimension | 1.36 (0.09) | 1.36 (0.07)
Statistical Analysis 1: Comparison: Baseline vs 7 Months; Test type: Superiority; p = 0.37, t-test, 2 sided

4. Secondary Outcome: Increase in Peak Oxygen Consumption on Cardiopulmonary Exercise Testing After Training
Description: peak oxygen consumption measured by cardiopulmonary exercise testing on a semi-recumbent cycle ergometer. Reported standardised to age, gender, height and weight in ml/kg/min
Time Frame: Baseline and 7 months
Population: Three subjects did not have complete cardiopulmonary exercise testing results post marathon, two due to injuries sustained and one due to equipment failure.
  68 Participants underwent the cardiopulmonary exercise test at baseline but 65 Participants underwent the cardiopulmonary exercise test at 7 months.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Baseline | 7 Months
Number analyzed (Participants) | 68 | 65
ml/kg/min | 37.9 (6.3) | 38.4 (6.9)

5. Other Pre Specified Outcome: Change in NTproBNP Levels
Description: Serum biomarker level.
  No outcome data reported as during the conduct of the study remodelling was not seen from baseline to post-marathon study time-points and therefore NTproBNP levels were expected to remain unchanged and would not provide any additional value in the study and so was not undertaken.
Time Frame: Baseline and 7 months
Population: As no changes in remodelling data were demonstrated in the primary analysis, it was felt by the primary supervisor that NTproBNP levels would not be expected to change and further investigation and expense would not be of value. The initial hypothesis that NTproBNP levels would change was predicated on the assumption that remodelling changes would be found and correlation with biomarker elevation would have yielded some insights had remodelling occurred.
Arm/Group | Baseline | 7 Months
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes